CLINICAL TRIAL: NCT03652324
Title: Comparison of General Anesthesia and Deep Sedation in Enbronchial Coil Treatment
Brief Title: What Should be the Anesthesia Method in Endobronchial Coil Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Collaborators: Bozok University (Other)
Responsible Party: Principal Investigator, Gamze Talih, Doctor, Bozok University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 60174989-23
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Coil Treatment; Deep Sedation
Keywords: coil treatment; general anesthesia; deep sedation
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- randomized (Other)
  Interventions: Other: method

INTERVENTIONS:
Other: method — to compare the use of general anesthesia and deep sedation

SUMMARY:
This prospective, randomize study was conducted in a university hospital. Bronchoscopic lung volume reduction (BLVR) coil treatment has recently been introduced into clinical practice as an alternative for patients chronic obstructive pulmonary disease (COPD) with severe refractory heterorogenous emphysema to conventional medical treatment. Thirty two patients diagnosed with (COPD) with severe refractory heterorogenous emphysema undergoing BLVR coil treatment were included in the study. Seventeen procedure were performed under general anesthesia and fifteen procedure were performed under deep sedation-analgesia. in the general anesthesia group peak pressure, air leakage and end-tidal carbon dioxide were recorded. In the both groups pulse oximeter, transcutaneous carbondioxide, recovery time, bronchospasm, laryngospasm, pneumothorax, massive bleeding were recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with COPD with undergoing BLVR coil treatment.

Exclusion Criteria:

* patients who refuse to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
recovery time measurement | 2 hours
  to compare the recovery time in both groups
complication rate | 2 hours
  to compare the complication rate in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Bozok University, Yozgat, Eyalet/Yerleşke, Turkey (Türkiye)